CLINICAL TRIAL: NCT01184014
Title: Hospital Insulin Protocol Aims for Glucose Control in Corticosteroid-induced Hyperglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04000-10-C
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Results first posted 2013-11-18 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2013-11

CONDITIONS: Hyperglycemia
Keywords: corticosteroid; hyperglycemia; hospital; corticosteroid induced hyperglycemia in the hospital
MeSH Terms: conditions — Hyperglycemia | interventions — Insulin, Isophane; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): a study-specific steroid (NPH) dosing algorithm plus standard recommended care. The intervention is Neutral Protamine Hagedorn (NPH) insulin plus complete insulin orders (CIO).
  Interventions: Drug: NPH insulin plus Complete Insulin Orders
- Control group (Active Comparator): the standard recommended care (Methodist Hospital Complete Insulin Orders)
  Interventions: Drug: Complete Insulin Orders

INTERVENTIONS:
Drug: NPH insulin plus Complete Insulin Orders — NPH dosed per study-specific algorithm which incorporates total daily dosage of steroid to determine NPH dose. Complete insulin orders include background, meal-time and correction factor.
  Other Names: lantus; glargine; humalog; lispro
  Arms: Experimental group
Drug: Complete Insulin Orders — 3-part insulin which includes background, meal-time and correction factor
  Other Names: lantus; glargine; humalog; lispro
  Arms: Control group

SUMMARY:
The objective of this study is to determine the best insulin regimen for hospitalized patients who receive high doses of steroids who have high blood glucose.

DETAILED DESCRIPTION:
The overall study objective of this research is to establish the efficacy and assure the safety of achieving glycemic control in hospitalized patients who receive greater than physiologic doses of steroids. This study will compare 2 methods of achieving glycemic control in hospitalized patients who develop steroid-induced hyperglycemia (blood glucose (BG) >180 mg/dL): 1) a study-specific steroid NPH dosing algorithm plus standard recommended care (Experimental group) vs. 2) the standard recommended care (Methodist Hospital Complete Insulin Orders (Control group).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years who receive steroids in doses greater than physiologic replacement levels of ≥ 10 mg Prednisone or its equivalent of dexamethasone or methylprednisolone.
* Have signed the consent form for the study
* Have a BG > 180 mg/dL any time during the first 24 hour of steroid administration that is above physiological replacement ( ≥ 10 mg Prednisone or equivalent)
* Are scheduled to be in hospital ≥ 2 days.

Exclusion Criteria:

* Unable to read or understand English
* History of psychiatric disability affecting informed consent or compliance with drug intake
* Type 1 diabetes
* Acute or chronic renal failure (creatinine clearance < 30 mL/min estimated by method of Cockcroft and Gault)
* Patients in Hospice Care
* Age <18 years
* Previously enrolled in this study.
* Not appropriate for the steroid protocol in judgment of the principal investigator and/or attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- Park Nicollet Health Services Methodist Hospital, Saint Louis Park, Minnesota, United States

REFERENCES:
- [Background] Clore JN, Thurby-Hay L. Glucocorticoid-induced hyperglycemia. Endocr Pract. 2009 Jul-Aug;15(5):469-74. doi: 10.4158/EP08331.RAR. PMID 19454391
- [Background] Derendorf H, Hochhaus G, Mollmann H, Barth J, Krieg M, Tunn S, Mollmann C. Receptor-based pharmacokinetic-pharmacodynamic analysis of corticosteroids. J Clin Pharmacol. 1993 Feb;33(2):115-23. doi: 10.1002/j.1552-4604.1993.tb03930.x. PMID 8440759
- [Background] Donihi AC, Raval D, Saul M, Korytkowski MT, DeVita MA. Prevalence and predictors of corticosteroid-related hyperglycemia in hospitalized patients. Endocr Pract. 2006 Jul-Aug;12(4):358-62. doi: 10.4158/EP.12.4.358. PMID 16901792
- [Derived] Grommesh B, Lausch MJ, Vannelli AJ, Mullen DM, Bergenstal RM, Richter SA, Fish LH. HOSPITAL INSULIN PROTOCOL AIMS FOR GLUCOSE CONTROL IN GLUCOCORTICOID-INDUCED HYPERGLYCEMIA. Endocr Pract. 2016 Feb;22(2):180-9. doi: 10.4158/EP15818.OR. Epub 2015 Oct 22. PMID 26492541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from May 2011 to August 2012. Location: Hospital.
Groups:
- Experimental Group: a study-specific steroid NPH dosing algorithm plus standard recommended care
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 35 | 37
Completed | 30 | 31
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 35 | 37 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (14.2) | 71.6 (44.6) | 69.4 (33.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 35 | 37 | 72

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Glucose of All Readings
Description: Starting 3 hours after the initial index blood glucose (BG) >180 measure, across the entire hospital stay or up through 5 days if hospital length of stay (LOS) is > 5 days
Time Frame: starting 3 hours after the initial index BG>180 measure, across the entire hospital stay or up through 5 days if hospital LOS is > 5 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 30 | 31
mg/dL | 157.2 (6.1) | 181.8 (32.6)

ADVERSE EVENTS:
Time Frame: Adverse event data collected over complete length of inpatient stay, up through 5 days.
Description: All subjects glucose level tests were reviewed looking for incidence of severe hypoglycemia (< 50 mg/dL)
Arm/Group | Experimental Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes